CLINICAL TRIAL: NCT03829631
Title: Lumbar Brace Deployment in The Emergency Department for Benign Low Back Pain: Effectiveness and Impact on Pain, Spine Function, Analgesic Use and Community Resources
Brief Title: Lumbar Brace Deployment in the Emergency Department for Benign Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: American Orthotic and Prosthetic Association (Other); Curtin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00085904
Record Dates: First submitted 2019-01-24; First posted 2019-02-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain; Brace; Emergencies; Pain; Health Care Resources
MeSH Terms: conditions — Low Back Pain; Emergencies; Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, superiority, 1:1 parallel randomised control trial with concealed allocation. Superiority will be based on a minimally clinically significant difference of our primary outcome measure (Numerical Pain Rating Scale, a 0-10 point scale).
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of each intervention, blinding will not be feasible for participants. However, outcomes assessor and adjudicators, as well as the statistician, will be blinded to the actual allocation. The investigators will develop two interpretations of our results based on a blinded review of the primary outcome data (intervention A vs. intervention B). One scenario will assume intervention A was brace and the other will assume intervention A was routine recommendations. Only after our team has agreed that there will be no further changes in the interpretation of the scenarios will the randomisation code be broken, and the correct interpretation used in manuscript preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be instructed to follow their current low back pain management program, in addition, they will be instructed to wear a lumbar brace (Horizon 627 Lumbar Brace) during the day for four weeks only when they are in pain in addition to their current management program.
  Interventions: Device: Horizon 627 Lumbar Brace, Aspen Medical Company, Oak Canyon, Irvine, CA 92618
- Control (No Intervention): Participants will be instructed to follow their current low back pain management program.

INTERVENTIONS:
Device: Horizon 627 Lumbar Brace, Aspen Medical Company, Oak Canyon, Irvine, CA 92618 — The brace is an FDA Class I, one-size adjustable design to fit waists ranging from 24-70 inches. Participants will be instructed to wear the brace for six weeks during the daytime
  Arms: Intervention

SUMMARY:
Low back pain accounts for billions of dollars in health care expenditures. Most cases of back pain do not have a clear cause. Thus, low back pain management methods usually rely on targeting people' pain and discomfort. Painkillers, including opioids, are usually prescribed in the emergency departments for people with low back pain. But, like all medications, painkillers can have side effects, and some of those can be serious. There are also serious concerns about the overuse of painkillers. Thus, newer pain management methods are needed to reduce the use of painkillers in people with low back pain. Lumbar braces are one of the underutilized low back pain management methods in the emergency departments. Like crutches for leg and ankle injuries, they can minimise movements of the spine. This may decrease people pain and improve their function. This may also reduce the use of painkillers. In support of this approach, two recent studies conducted in a primary-care setting observed a reduction in the use of painkillers in people with low back pain who wore lumbar braces. The investigators are conducting this study to determine if wearing a lumbar brace for 4 weeks following emergency department presentation will reduce people's pain and discomfort and increase spine function. This may decrease the use of painkiller and future use of healthcare resources. This research study may also assist emergency-department staff with offering new recommendations to improve the quality of clinical decisions.

DETAILED DESCRIPTION:
BACKGROUND/SIGNIFICANCE

The global point prevalence of activity-limiting low back pain was 7.3% in 2015, implying that 540 million people were affected at one time. Although people with acute or chronic low back pain usually improve in the first six weeks, they usually suffer from low to moderate levels of pain and disability in the first year. Low back pain is an urgent global public health concern, accounting for billions of dollars in health care expenditures. Much of this spending is for high-cost, low-value care such as evaluating low back pain in the emergency department; only 3% of persons with low back pain attending the emergency department are admitted to the hospital while those who are discharged leave without effective pain control. This low-value approach is thought to increase use of additional health-related resources including repeat use of the emergency department for future low back pain complaints and use of opioids. This reduces limited available resources that should more appropriately be used for other health care needs.

While emergency departments routinely recommend analgesics for low back pain (paracetamol, nonsteroidal anti-inflammatory drugs, opioids, etc.), current guidelines do not support this approach; only nonsteroidal anti-inflammatory drugs are recommended as second-line/adjunctive treatment. As such, there is a critical need to provide emergency-department staff with better short-term pain control solutions. One underutilized pain-control solution in emergency departments is lumbar orthoses. Like crutches for leg or ankle injuries, lumbar orthoses can minimise lumbar spine movements, which can reduce pain and discomfort while preserving important aspects of daily function. In support of this approach, two recent randomised controlled trials conducted in a primary-care setting observed a reduced analgesic consumption in low back pain patients who received lumbar orthoses.

HYPOTHESES

1. Wearing a semi-rigid lumbar brace for 4 weeks following emergency department presentation will reduce participant pain and discomfort;
2. The same bracing protocol will improve spine function;
3. The same bracing protocol will decrease analgesic consumption including opioids;
4. The same bracing protocol will decrease future use of healthcare resources.

SPECIFIC AIMS

1. PRIMARY: To determine if lumbar bracing for 30 days after the emergency department presentation will reduce low back pain;
2. SECONDARY: To determine if this same bracing protocol will improve spinal function and quality of life;
3. SECONDARY: To establish if this same bracing protocol will reduce prescription and/or consumption of analgesics;
4. EXPLORATORY: To establish if this same bracing protocol will reduce back pain-related use of health resources (e.g., emergency department, primary care, imaging, and non-prescription management).

RESEARCH PLAN

Study Design

This project is a prospective, superiority, 1:1 allocation, randomised controlled trial with concealed allocation. Specifically, the investigators will recruit people with benign low back pain presenting to the Emergency Department. Superiority will be based on a minimally clinically significant difference of our primary outcome measure (Numerical Pain Rating Scale, a 0-10-point scale). Statisticians will be blinded to group allocation. The investigators will exclude those with a confirmed cause of low back pain (e.g. trauma), significant compression of the spinal cord/nerves and on-going workers' compensation or litigation cases.

Procedure

After obtaining approval from the University of Alberta's Health Research Ethics Board, the investigators will invite people with benign low back pain presenting to Emergency Department (to be determined) to consent and take part in the study. After enrolment, each participant will be given a study number to maintain and track her/his records. The participant will be then provided with a Research Electronic Data Capture (REDCap) secure web address to complete various data collection surveys (e.g. demographics).

Baseline session

The investigators will collect demographics, comorbidities, medication, and self-reported histories of imaging and treatment. Participants will use self-reported outcome tools to quantify pain (Numerical Pain Rating Scale) and function (Roland-Morris Disability Questionnaire). The investigators will then randomize participants to one of two arms: brace or no brace.

All participants will be instructed that the current study will not substitute their current back pain management program. Participants in the intervention arm will be fitted with a semi-rigid prefabricated lumbar brace (Horizon 627 Lumbar Brace, Aspen Medical Company, Oak Canyon, Irvine, CA 92618). The brace is a one-size adjustable design to fit waists ranging from 24-70 inches. Participants will be instructed to wear the brace for six weeks. As this brace is semi-rigid, it does not prevent motion - only reduces motion in the lumbar areas. Our prior work and that of others have shown that this type of bracing does not reduce spinal function and is not associated with atrophy.

Randomisation: the investigators will deploy the REDCap randomisation tool to assign participants evenly into the intervention and control groups. The tool uses a defined parameter (subject ID in this study) to create a template allocation table. The on-site research assistant will enter each participant's REDCap record and then click the "Randomize" button. This will trigger REDCap to check the allocation table and display the group to which the participant should be assigned. The assignment is permanent and not editable within the participant record and, like all other activity within REDCap, is tracked and not modifiable in the audit log.

Self-reported questionnaires: the investigators will measure participants' pain level using the Numeric Pain Rating Scale. the investigators will use the Roland-Morris Disability Questionnaire and the Oswestry Disability Index to measure participant function and disability level.

Immediately after wearing the brace (only the intervention group): To assess the immediate impact of the brace, participants will use self-reported outcome tools on the REDCap to quantify pain (Numeric Pain Rating Scale) immediately after wearing the brace.

To measure the quality (how tightly the brace has been worn) and quantity (how much time the brace has been worn) of brace usage, a low-powered portable heat and load monitoring system will be embedded within the pressure pad of the brace. The force measurement part of the monitoring system is sensitive to the forces normal to the brace surface, but not to shear forces, and can be deployed to monitor the quality of the brace wear by participants.28 The temperature part of the monitoring system gives an accurate and stable output over the temperature range from 5 °C to 50 °C,29 and can be deployed to monitor how long the brace has been worn during the brace treatment.

Follow-up (both groups)

All participants will receive a series of short message service (SMS) text messages 3 times/week for 4 weeks to evaluate Numerical Pain Rating Scale, Roland-Morris Disability Questionnaire, brace usage, and analgesic consumption. The investigators will also collect a series of outcomes and interview questions by SMS at 2 and 3 months.

The end of the enrollment

The investigators will use participant healthcare numbers (obtained at baseline with consent) to perform an exploratory analysis through the Alberta Bone and Joint Health Network of health care resource utilization in the year before and during the trial (e.g. prescriptions filled, primary care or emergency department visits, imaging usage, etc.).

ANALYSIS METHODS

Blinding

Due to the nature of each intervention, blinding will not be feasible for participants. However, the outcomes assessor, outcome adjudicators, and the statistician will be blinded to the actual allocation. The investigators will develop two interpretations of our results based on a blinded review of the primary outcome data (intervention A vs. intervention B). One scenario will assume intervention A was brace and the other will assume intervention A was routine recommendations. Only after our team has agreed that there will be no further changes in the interpretation of the scenarios will the randomisation code be broken, and the correct interpretation used in manuscript preparation.

Statistical Analysis

The investigators will employ a repeated model of analysis of variance to compare pain level between groups. The investigators will use age, gender, and pain severity as potential covariates if randomization does not result in group equivalence. The investigators will also estimate the effect size of differences between and within the groups for pain using Cohen's d.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Ambulatory
* Able to read and understand English
* Living in Edmonton
* Presenting to an emergency department

Exclusion Criteria:

* Back pain due to systemic or specific disease such as known cancer, spinal infection, fracture, or ankylosing spondylitis
* Pregnancy
* Significant compression of the spinal cord/nerves
* Previous back surgery
* On-going workers' compensation or litigation cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the pain level | Week 6
  The change in the pain level between the baseline and 6-week follow-up will be evaluated using the Numeric Pain Rating Scale [0-10]. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing the "worst pain imaginable".
Change in the pain level | Month 4
  The change in the pain level between the baseline and 4-month follow-up will be evaluated using the Numeric Pain Rating Scale [0-10]. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing the "worst pain imaginable".
Change in the pain level | Month 8
  The change in the pain level between the baseline and 8-month follow-up will be evaluated using the Numeric Pain Rating Scale [0-10]. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing the "worst pain imaginable".
Change in the pain level | Month 12
  The change in the pain level between the baseline and 12-month follow-up will be evaluated using the Numeric Pain Rating Scale [0-10]. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing the "worst pain imaginable".

SECONDARY OUTCOMES:
Change in the self-reported disability level - Questionnaire A | Week 6
  The change in the self-reported disability between the baseline and 6-week follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported disability level - Questionnaire A | Month 4
  The change in the self-reported disability between the baseline and 4-month follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported disability level - Questionnaire A | Month 8
  The change in the self-reported disability between the baseline and 8-month follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported disability level - Questionnaire A | Month 12
  The change in the self-reported disability between the baseline and 12-month follow-up will be evaluated using the Oswestry Disability Index [0-100 scale].
Change in the self-reported disability level - Questionnaire B | Week 6
  The change in the self-reported disability between the baseline and 6-week follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale].
Change in the self-reported disability level - Questionnaire B | Month 4
  The change in the self-reported disability between the baseline and 4-month follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale].
Change in the self-reported disability level - Questionnaire B | Month 8
  The change in the self-reported disability between the baseline and 8-month follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale].
Change in the self-reported disability level - Questionnaire B | Month 12
  The change in the self-reported disability between the baseline and 12-month follow-up will be evaluated using the Roland-Morris Low Back Pain and Disability Questionnaire Index [0-24 scale].

OTHER OUTCOMES:
Change in healthcare resource utilization- regulated prescriptions filled (after enrollment) | Month 12
  The change in healthcare resource utilization, measured by counting the number of back-pain related regulated prescriptions filled from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- primary care visits (after enrollment) | Month 12
  The change in healthcare resource utilization, measured by counting the number of back-pain related primary care visits from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- specialist visits (after enrollment) | Month 12
  The change in healthcare resource utilization, measured by counting the number of back-pain related specialist visits from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- imaging (after enrollment) | Month 12
  The change in healthcare resource utilization, measured by counting the number of back-pain related imaging from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- allied health visits (after enrollment) | Month 12
  The change in healthcare resource utilization, measured by counting the number of back-pain related allied health visits from the baseline and the past 12 months after enrollment
Change in healthcare resource utilization- regulated prescriptions filled (before enrollment) | 12 Month
  The change in healthcare resource utilization, measured by counting the number of back-pain related regulated prescriptions filled from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- primary care visits (before enrollment) | 12 Month
  The change in healthcare resource utilization, measured by counting the number of back-pain related primary care visits from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- specialist visits (before enrollment) | 12 Month
  The change in healthcare resource utilization, measured by counting the number of back-pain related specialist visits from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- imaging (before enrollment) | 12 Month
  The change in healthcare resource utilization, measured by counting the number of back-pain related imaging from the past 12 months before enrollment and baseline.
Change in healthcare resource utilization- allied health visits (before enrollment) | 12 Month
  The change in healthcare resource utilization, measured by counting the number of back-pain related allied health visits from the past 12 months before enrollment and baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Vahid Abdollah, PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Perth Hospital, Perth, Australia

IPD SHARING:
Plan to Share IPD: No